CLINICAL TRIAL: NCT00734019
Title: A Prospective, Non-comparative, Multicentre, Multinational Study to Determine the Survivorship of the P.F.C. Fixed Bearing Knee System Using a Moderately Cross-linked Polyethylene Insert and a Cobalt Chrome Tibial Tray.
Brief Title: Survivorship of the Press Fit Condylar (P.F.C.) Sigma Fixed Bearing Knee With a Cobalt Chrome Tibial Tray
Status: Completed | Type: Observational
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Other Study IDs: CT 04/16
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee, TKR, PFC Sigma
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- P.F.C. Sigma Knee System: Orthopaedic implant for primary total knee replacement with a cobalt-chrome tibial tray and a moderately cross-linked polyethylene tibial insert
  Interventions: Device: P.F.C. Sigma Knee

INTERVENTIONS:
Device: P.F.C. Sigma Knee — Orthopaedic implant for primary total knee replacement with a cobalt-chrome tibial tray and a moderately cross-linked polyethylene tibial insert

SUMMARY:
The study will determine the survivorship of the fixed bearing P.F.C. Sigma knee with a cobalt chrome tibial tray at 5 years.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the survivorship of the P.F.C. fixed bearing knee system using a cobalt chrome tibial tray and moderately cross-linked polyethylene insert at 5-Years. The secondary objectives of this investigation are to evaluate additional clinical outcomes to provide further information on the performance of the P.F.C. fixed bearing knee system using a moderately cross-linked polyethylene insert and cobalt chrome tibial tray. These outcomes will include Radiographic assessment, American Knee Society Score, Oxford Knee Score and SF-12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have given voluntary written informed consent to participate in this study
* Subjects for whom primary total knee replacement is indicated due to degenerative joint disease, including rheumatoid arthritis, osteoarthritis, avascular necrosis, and post traumatic arthritis, which is causing pain, deformity, or limitation of function uncontrolled by medical treatment.
* Subjects who, in the opinion of the Investigator, are able to understand this study, co-operate with the investigational procedures and are willing to return to the hospital for all scheduled post-operative follow ups.
* Male or Female subjects who are skeletally mature and for whom an appropriate size of device is available
* The following subjects are not considered eligible and must not be recruited to the investigation

Exclusion Criteria:

* Subjects scheduled for revision total knee arthroplasty, or who have had previous surgery to their knee except menisectomy, arthroscopy or synovectomy.
* Subjects aged over 80 Years
* Subjects experiencing any condition that may, in the opinion of the investigator, interfere with the total knee replacements survival or outcome (e.g. Pagets disease, Charcots disease, severe osteoporosis etc).
* Subjects who have evidence of active infections, which may spread, to other areas of the body (e.g. osteomyelitis, pyrogenic infection of the knee joint, overt infection etc)
* Subjects who are currently participating in any other clinical investigation of a device or pharmaceutical.
* Subjects having non-contained defects in the tibia or femur necessitating bone graft.
* Subjects with psychosocial disorders that would limit rehabilitation
* Subjects with a known history of poor compliance to medical treatment
* Subjects who are known drug or alcohol abusers.
* Other contraindications for the use of the P.F.C. ® S fixed bearing knee system as listed in the package insert.
* Women who are pregnant
* Subjects who are currently involved in any injury litigation claims

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2005-10-01 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a survivorship analysis of the P.F.C. fixed bearing knee system with a cobalt chrome tibial tray and moderately cross linked polyethylene insert at the five-year time point. | 5 years

SECONDARY OUTCOMES:
Changes from pre-operative assessment Clinical outcome and patient-derived outcome in terms of joint-specific quality of life. | 3 month, 1,3, 5 and 10 years

CONTACTS AND LOCATIONS:
Locations (5):
- Asklepios Klinic/ Lindenlohe Orthopeadic Hospital, Schwandorf in Bayern, Deutschland, Germany
- Hospital S Antonìo Of Padova, Padua, Italy
- United Kingdom (3):
  - Princess Alexandra Hospital, Harlow, Essex
  - Queen Margaret Hospital, Dunfermline, Fife
  - Arrowe Park Hospital, The Wirral, Merseyside